CLINICAL TRIAL: NCT03827499
Title: Effects of β-hydroxy-β-methylbutyrate (HMB) Supplementation in Addition to Multicomponent Exercise in Old Adults Living in Nursing Homes
Brief Title: HMB Supplementation in Addition to Multicomponent Exercise in Old Adults
Acronym: HEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Javier Courel Ibáñez, Ph.D, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2131/2018
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Aging; Frail Elderly Syndrome; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ex-HMB (Experimental): HMB dietary supplementation and Multicomponent physical exercise program
  Interventions: Dietary Supplement: HMB dietary supplementation; Other: Multicomponent physical exercise program
- NoEx-HMB (Experimental): HMB Dietary supplementation
  Interventions: Dietary Supplement: HMB dietary supplementation
- Ex-Plac (Placebo Comparator): Multicomponent physical exercise program
  Interventions: Other: Multicomponent physical exercise program
- Controls (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: HMB dietary supplementation — Intervention groups including HMB supplementation (Ex-HMB and NoEx-HMB) will receive a 3 g daily dose of free acid HMB in powder form dissolved freely into 250 mL of water during a 24-week intervention
  Arms: Ex-HMB; NoEx-HMB
Other: Multicomponent physical exercise program — Intervention groups including exercise (Ex-HMB and Ex-Plac) will complete an individualized multicomponent training program, five days a week during 24 weeks.
  Arms: Ex-HMB; Ex-Plac

SUMMARY:
Evidence supports the fact that multicomponent exercise and β-hydroxy-β-methylbutyrate (HMB) supplementation are, separately, effective in improving old adult's health and palliate functional metabolic diseases in the elderly. However, the true effect of HMB supplementation combined with a tailored exercise program in frail old adults is still unknown. Thus, the aim of the HEAL study is to assess the effects of the combination of a daily multicomponent exercise and resistance training intervention in addition to HMB supplementation on old adults' health.

DETAILED DESCRIPTION:
Evidence supports the fact that multicomponent exercise and β-hydroxy-β-methylbutyrate (HMB) supplementation are, separately, effective in improving old adult's health and palliate functional metabolic diseases in the elderly. However, the true effect of HMB supplementation combined with a tailored exercise program in frail old adults is still unknown.

Thus, the aim of the HEAL study is to assess the effects of the combination of a daily multicomponent exercise and resistance training intervention in addition to HMB supplementation on old adults' health.

The findings of the HEAL study will help professionals from public health systems to identify cost-effectiveness and innovative actions to improve older people's health and quality of life, and endorse exercise practice in older adults living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥70 years living in a nursing home
* Be able to follow an active physical rehabilitation program
* Be able to read and wright
* Voluntary participation
* Capable and willing to provide an informed consent

Exclusion Criteria:

* Acute heart attack (recent 3-6 months) or unstable angina
* Uncontrolled atrial or ventricular arrhythmias
* Aortic dissecting aneurysm
* Severe aortic stenosis
* Acute endocarditis / pericarditis
* Uncontrolled high blood pressure (>180/100 mmHg)
* Acute thromboembolism
* Acute or severe heart failure
* Acute or severe respiratory failure
* Uncontrolled postural hypotension
* Uncontrolled acute decompensated diabetes mellitus or low blood sugar
* A recent fracture in the last month.
* Coincident participation in any intervention trial
* HMB contraindication, intolerance, or allergy
* Community-dwelling people
* Have regularly performed exercise (>20 minutes >3 days/week) in the last 3 months
* Malignant diseases (exceptions: basal or squamous-cell skin carcinoma or carcinoma in situ of the uterine cervix)
* Revascularization within 1 year
* Severe loss of vision, hearing, or communicative ability
* Conditions preventing cooperation

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in physical functional performance based on the Short Physical Performance Battery (SPPB) score | Baseline to 25 Weeks
  Summary scores range from 0-12 and higher scores denote higher physical performance.

SECONDARY OUTCOMES:
Change in Handgrip strength (kg) | Baseline to 25 Weeks
  Using a dynamometer
Change in lower-body strength (kg) | Baseline to 25 Weeks
  Seated leg press one-repetition maximun test
Change in upper-body strength (kg) | Baseline to 25 Weeks
  Vertical bench press one-repetition maximun test
Change in lower-body strength power output (m/s) | Baseline to 25 Weeks
  Seated leg press load-velocity profile
Change in upper-body strength power output (m/s) | Baseline to 25 Weeks
  Vertical bench press load-velocity profile
Change in frailty (score) | Baseline to 25 Weeks
  Frailty phenotype determination using Fried's criteria
Change in lean body mass (kg) | Baseline to Week 25
  Change in lean body mass using dual energy x-ray absorptiometry
Change in lipid profile | Baseline to Week 25
  Plasma total, high-density lipoprotein and low-density lipoprotein cholesterol and triglycerides (all in mg/dL)
Change in glycaemic profile | Baseline to Week 25
  Plasma glucose, insulin and glycosylated haemoglobin (all in mg/dL)
Change in Thyroid-Stimulating Hormone (mIU/L) | Baseline to Week 25
Change in Disability (Lawton index scores) | Baseline to 25 Weeks
  Disability in instrumental activities of daily living.
Change in Disability (Barthel index scores) | Baseline to 25 Weeks
  Disability in basic activities of daily living
Change in Comorbidity (score) | Baseline to 25 Weeks
  When a participant presents two or more geriatric syndromes from a list of selected geriatric syndromes
Change in cognitive function (score) | Baseline to 25 Weeks
  Using the Mini-Mental State Examination
Change in depression (score) | Baseline to 25 Weeks
  Using the 15-item Yesavage geriatric depression

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Sciences, Murcia, San Javier, Spain

REFERENCES:
- [Derived] Courel-Ibanez J, Pallares JG; HEAL study group. Effects of beta-hydroxy-beta-methylbutyrate (HMB) supplementation in addition to multicomponent exercise in adults older than 70 years living in nursing homes, a cluster randomized placebo-controlled trial: the HEAL study protocol. BMC Geriatr. 2019 Jul 5;19(1):188. doi: 10.1186/s12877-019-1200-5. PMID 31277595